CLINICAL TRIAL: NCT00915759
Title: Sutureless Cryopreserved Amniotic Membrane Graft (ProKera) and Wound Healing After Photorefractive Keratectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: BioTissue Holdings, Inc (Industry); St. John's Hospital (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-6961
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Results first posted 2013-09-20 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Corneal Wound Healing
Keywords: ProKera; Amniotic membrane; Photorefractive Keratectomy; PRK; time to re-epithelialization

ARMS (2):
- ProKera (Active Comparator)
  Interventions: Device: ProKera
- Bandage contact lens (Placebo Comparator)
  Interventions: Device: Bandage contact lens

INTERVENTIONS:
Device: ProKera — ProKera placed in non-dominant eye after photorefractive keratectomy (PRK)
  Arms: ProKera
Device: Bandage contact lens — Bandage contact lens placed in dominant eye, the current standard after photorefractive keratectomy (PRK)
  Arms: Bandage contact lens

SUMMARY:
The purpose of this study is to evaluate the effect of ProKera on corneal wound healing after photorefractive keratectomy (PRK) in terms of re-epithelialization, pain, adverse effects, visual recovery, refractive accuracy, and corneal clarity.

ELIGIBILITY:
Inclusion Criteria:

* Active duty US Army Soldiers eligible for care at WRAMC.
* Male or female, of any race, and at least 21 years old at the time of the preoperative examination, and have signed and informed consent. The lower age limit of 21 years is intended to ensure documentation of refractive stability.
* Subject must expect to be located in the greater Washington, District of Columbia area for a 12 month period post-operatively.
* Consent of the subject's command (active duty) to participate in the study.
* Access to transportation to meet follow-up requirements.

Exclusion Criteria:

* Any reason to be excluded for PRK.
* Female subjects who are pregnant, breast-feeding or intend to become pregnant during the study. Female subjects will be give a urine pregnancy test prior to participating in the study to rule out pregnancy. [Pregnancy and breastfeeding are contraindications to refractive surgery in general, including PRK, whether participating in this study or not].
* Patients with known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course.
* Any physical or mental impairment that would preclude participation in any of the examinations.
* Anterior basement membrane dystrophy.
* History of recurrent epithelial erosion.
* Significant dry eye (symptomatic with Schirmer test < 5 mm at 5 minutes).
* Other corneal epithelial disorder or healing abnormality.
* Patients with unusually tight eyelids close to the eyeball making it difficult and/ or painful to insert anything (e.g., ProKera) between the eyelid and globe.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Stutzman, MD, Principal Investigator — WRNMMC
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ProKera/Bandage Contact Lens: Each patient received ProKera on dominant eye and bandage contact lens on fellow non-dominant eye after photorefractive keratectomy (PRK)
Period: Overall Study
Arm/Group | ProKera/Bandage Contact Lens
Started | 40 (number of participants)
Completed | 40 (number of participants)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- ProKera and Bandage Contact Lens: Each participant received ProKera on dominant eye and bandage contact lens on fellow non-dominant eye after PRK
Arm/Group | ProKera and Bandage Contact Lens
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Days to Complete Re-epithelialization
Description: measured as number of days to complete re-epithelialization, as assessed by daily examination using slit lamp biomicroscopy
Time Frame: participants will be followed daily until complete re-epithelialization, an expected average of 3-5 days post-operatively
Population: Each participant received ProKera on dominant eye and bandage contact lens on fellow non-dominant eye after PRK. For group 1, ProKera and bandage contact lens were left in place until complete corneal re-epithelialization (healing).
Measure: Mean (Standard Deviation); unit: days to complete re-epithelialization
Units Other Than Participants: eyes
Groups:
- ProKera: Group 1: ProKera in place until complete corneal re-epithelialization (healing)
- Bandage Contact Lens: Group 1: bandage contact lens in place until complete corneal re-epithelialization (healing)
Arm/Group | ProKera | Bandage Contact Lens
Number analyzed (Participants) | 9 | 9
Number analyzed (eyes) | 9 | 9
days to complete re-epithelialization | 4.6 (1.6) | 4.1 (1.4)

2. Primary Outcome: Number of Days to Complete Re-epithelialization
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Each participant received ProKera on dominant eye and bandage contact lens on fellow non-dominant eye after PRK.For group 2, ProKera and bandage contact lens were left in place until postoperative day 3.
Measure: Mean (Standard Deviation); unit: days to complete re-epithelialization
Units Other Than Participants: eyes
Groups:
- ProKera: Group 2: ProKera in place until postoperative day 3
- Bandage Contact Lens: Group 2: bandage contact lens in place until postoperative day 3
Arm/Group | ProKera | Bandage Contact Lens
Number analyzed (Participants) | 15 | 15
Number analyzed (eyes) | 15 | 15
days to complete re-epithelialization | 5.2 (3.5) | 3.9 (1.1)

3. Primary Outcome: Number of Days to Complete Re-epithelialization
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Each participant received ProKera on dominant eye and bandage contact lens on fellow non-dominant eye after PRK.For group 3, ProKera and bandage contact lens were left in place until postoperative day 1.
Measure: Mean (Standard Deviation); unit: days to complete re-epithelialization
Units Other Than Participants: eyes
Groups:
- ProKera: Group 3: ProKera in place until postoperative day 1
- Bandage Contact Lens: Group 3: bandage contact lens in place until postoperative day 1
Arm/Group | ProKera | Bandage Contact Lens
Number analyzed (Participants) | 16 | 16
Number analyzed (eyes) | 16 | 16
days to complete re-epithelialization | 4.0 (0.8) | 3.8 (0.5)

4. Secondary Outcome: Post-operative Pain Score Ranging From 0 (None) to 10 (Worst Possible Pain)
Description: measured subjectively using the Visual Analog Scale (VAS) ranging from 0 (none) to 10 (worst possible pain)
Time Frame: Day 1
Population: eyes
Measure: Mean (Standard Deviation); unit: VAS score
Units Other Than Participants: eyes
Groups:
- ProKera: ProKera: ProKera placed in non-dominant eye after PRK
- Bandage Contact Lens: Bandage contact lens: Bandage contact lens placed in dominant eye, the current standard after PRK
Arm/Group | ProKera | Bandage Contact Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (eyes) | 40 | 40
VAS score | 4.6 (3.3) | 4.8 (2.5)

5. Secondary Outcome: Number of Eyes With Complications/Adverse Events
Time Frame: up to one year post-operatively
Population: eyes
Measure: Count of Units; unit: eye
Units Other Than Participants: eye
Arm/Group | ProKera | Bandage Contact Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (eye) | 40 | 40
eye
  Spontaneous extrusion of the graft (or BCL) at first postop week | 1 | 0
  Delayed epithelial healing in early postop | 1 | 0
  Persistent epithelial defect in early postop | 2 | 0
  Corneal infiltrates (inflammatory) in early postop | 4 | 4
  non-granulomatous anterior uveitis at 1 week postop | 1 | 0

6. Secondary Outcome: Number of Eyes Achieving Uncorrected Distance Visual Acuity of 20/20 or Better at 12 Months Post-operatively
Description: Uncorrected Distance Visual Acuity
Time Frame: one year post-operatively
Population: eyes
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | ProKera | Bandage Contact Lens
Number analyzed (Participants) | 35 | 35
Number analyzed (eyes) | 35 | 35
eyes | 34 | 35

7. Secondary Outcome: Number of Eyes With Manifest Spherical Equivalent Within +/- 0.50 Diopters of Emmetropia at 12 Months Post-operatively
Description: Manifest spherical equivalent within +/- 0.50 diopters of emmetropia
Time Frame: one year post-operatively
Population: eyes
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | ProKera | Bandage Contact Lens
Number analyzed (Participants) | 35 | 35
Number analyzed (eyes) | 35 | 35
eyes | 32 | 30

8. Secondary Outcome: Number of Eyes With Clinically Significant Corneal Haze
Description: clinically significant corneal haze (grade 2 or higher)
Time Frame: one year postoperatively
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | ProKera | Bandage Contact Lens
Number analyzed (Participants) | 35 | 35
Number analyzed (eyes) | 35 | 35
eyes | 0 | 0

9. Secondary Outcome: Tear Total Protein Levels
Description: total protein levels
Time Frame: 1 month post-operatively
Population: samples
Measure: Mean (Standard Deviation); unit: mg/ml
Units Other Than Participants: samples
Arm/Group | ProKera | Bandage Contact Lens
Number analyzed (Participants) | 16 | 13
Number analyzed (samples) | 16 | 13
mg/ml | 9.6 (0.9) | 9.9 (0.8)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- ProKera; Bandage Contact Lens: Each patient received ProKera on dominant eye and bandage contact lens on fellow non-dominant eye after PRK
Arm/Group | ProKera | Bandage Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 9/40 | 4/40
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ProKera (N=40) | Bandage Contact Lens (N=40)
Acute non-granulomatous anterior uveitis (Eye disorders) | 1 (1) | 0 (0) — Acute, non-granulomatous anterior uveitis is a common, idiopathic inflammatory process that afflicts the iris and ciliary body.
Spontaneous extrusion of the graft (or BCL) at first postop week (Eye disorders) | 1 (1) | 0 (0)
Delayed epithelial healing in early postop (Eye disorders) | 1 (1) | 0 (0)
Persistent epithelial defect in early postop (Eye disorders) | 2 (2) | 0 (0)
corneal infiltrates (inflammatory) in early postop (Eye disorders) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other